CLINICAL TRIAL: NCT02609438
Title: The Effects of Short, Frequent Breaks in Sitting Versus Longer, Planned Breaks in Sitting on Sedentary Behavior and Metabolic Health Among Inactive Females Working Sedentary Jobs
Brief Title: An Intervention to Reduce Sitting Time at Work: Effects on Metabolic Health and Inactivity
Acronym: Up4Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Responsible Party: Principal Investigator, Emily Mailey, Assistant Professor, Kansas State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USRG-3046
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Sedentary Lifestyle
Keywords: worksite; intervention; sitting
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short breaks (Active Comparator): Participants instructed to stand/move for 1-2 minutes every half hour throughout the workday
  Interventions: Behavioral: Short breaks
- Long breaks (Active Comparator): Participants instructed to take two 15-minute activity breaks during each workday
  Interventions: Behavioral: Long breaks

INTERVENTIONS:
Behavioral: Short breaks — Following baseline testing, participants will attend a 30-minute individual orientation session, during which they will complete a planning worksheet with a research assistant. They will identify specific strategies they will use to accomplish the pre-specified goal (i.e., to take a 1-minute active break every 30 minutes during the workday). They will also identify potential barriers they will face and devise strategies for overcoming them. The intervention will officially start the Monday after the orientation session and will last for 8 weeks. Participants will receive a weekly email containing tips related to reducing sitting time at work. All participants will complete daily activity logs indicating the time and duration of all breaks from sitting across the 8-week intervention.
  Other Names: Up4Health - short breaks
  Arms: Short breaks
Behavioral: Long breaks — Following baseline testing, participants will attend a 30-minute individual orientation session, during which they will complete a planning worksheet with a research assistant. They will identify specific strategies they will use to accomplish the pre-specified goal (i.e., to take two 15-minute activity breaks during each workday). They will also identify potential barriers they will face and devise strategies for overcoming them. The intervention will officially start the Monday after the orientation session and will last for 8 weeks. Participants will receive a weekly email containing tips related to reducing sitting time at work. All participants will complete daily activity logs indicating the time and duration of all breaks from sitting across the 8-week intervention.
  Other Names: Up4Health - long breaks
  Arms: Long breaks

SUMMARY:
The purpose of this study is to determine whether varying the frequency and length of activity breaks during the workday will differentially impact sedentary behavior and health outcomes. Participants will be randomly assigned to take short, frequent breaks (i.e., 1 minute every half hour) or longer, planned breaks (i.e., two 15-minute walks) from sitting during the workday. They will be instructed to follow the assigned protocols for an 8-week intervention and the effects of their participation on sedentary behavior and a variety of health outcomes will be assessed. The investigators anticipate participants in both intervention arms will demonstrate significant reductions in daily sitting time, bit do not have an a priori hypothesis regarding the relative effectiveness of each approach.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether varying the frequency and length of activity breaks during the workday will differentially impact sedentary behavior and health outcomes. Women aged 25-50 who work full-time in sedentary jobs and participate in less than 60 minutes of overall physical activity per week will be recruited. At the beginning of the study participants will visit the laboratory to complete baseline health assessments and meet with a research assistant to outline their plan for reducing sitting time at work. At this time they will be randomly assigned to one of two groups: 1) Group A will be asked to take two 15-minute walks during each workday, or 2) Group B will be asked to stand up and move around for 1-2 minutes every half hour throughout the workday. The total duration of this program will be eight weeks. During this time participants will be asked to keep a brief daily log of their activity breaks during the workday. At the end of the 8-week program participants will return to the laboratory to repeat the health assessments.

ASSESSMENTS:

All participants will complete the following tests and procedures:

* Metabolic blood panel. Blood will be drawn from a quick finger stick to assess total cholesterol, triglycerides, LDL, HDL, and fasting glucose.
* DEXA scan. Participants will lie down on a body scanner for about 10 minutes to assess body composition.
* Body measurements. A trained research assistant will measure height, weight, and waist circumference.
* Blood pressure. A trained research assistant will measure blood pressure using an automated blood pressure cuff.

In addition, participants will complete the following assessments outside of the laboratory:

* Questionnaires: Participants will be asked to complete a series of questionnaires. This should take 15-20 minutes.
* Accelerometer: Participants will be asked to wear a motion sensor for a total of 21 days (three 7-day periods). This small apparatus is worn around the waist during the day. Participants will complete a log indicating when they were wearing the accelerometer each day.
* Food diary: Participants will be asked to record their food intake for a total of 9 days (three 3-day periods).

ELIGIBILITY:
Inclusion Criteria:

1. Work at least 35 hours per week
2. Spend at least 80% of working hours sitting (self-reported)
3. Engage in less than 60 minutes per week of leisure-time exercise (self-reported)
4. Not pregnant or planning to become pregnant in the next 3 months
5. Not currently trying to change weight
6. Speak English
7. Able to attend assessments
8. Willing to wear accelerometer
9. No anticipated significant conflicts during 8-week intervention

Exclusion Criteria:

1. Male
2. Working less than 35 hours per week
3. Spend >25% of working hours standing or active
4. Engage in more than 60 minutes per week of leisure-time exercise
5. Pregnant
6. Actively dieting or attempting to change weight

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in sedentary behavior during the workday | Baseline - week 8
  Measured by GT3X accelerometer

SECONDARY OUTCOMES:
Change in weight | Baseline - week 9
Change in blood pressure | Baseline - week 9
Change in resting heart rate | Baseline - week 9
Change in total cholesterol, HDL cholesterol, LDL cholesterol | Baseline - week 9
Change in triglycerides | Baseline - week 9
Change in fasting blood glucose | Baseline - week 9
Change in waist circumference | Baseline - week 9
Change in body composition | Baseline - week 9
  DEXA or bioelectrical impedance
Change in energy, tiredness, tension, and calmness | Baseline - week 8
  Activation-Deactivation Checklist
Change in fatigue severity, interference, and duration | Baseline - week 8
  Fatigue Symptom Inventory
Change in mood | Baseline - week 8
  Positive and Negative Affect Scale
Change in overall self-reported physical activity | Baseline - week 8
  International Physical Activity Questionnaire
Change in overall objectively measured physical activity | Baseline - week 8
  Measured by GT3X accelerometer
Change in diet quantity | Baseline - week 8
  Measured by 3-day food diary
Change in diet quality | Baseline - week 8
  Dietary Screener Questionnaire
Adherence to assigned protocols | up to 8 weeks
  Measured by activity logs

CONTACTS AND LOCATIONS:
Overall Officials: Emily L Mailey, PhD, Principal Investigator — Kansas State University

REFERENCES:
- [Derived] Casey K, Mailey EL, Rosenkranz RR, Swank A, Ablah E, Rosenkranz SK. Does dietary intake change during an intervention to reduce sedentary behavior and cardiovascular disease risk? A randomized comparative effectiveness trial. BMC Nutr. 2018 Apr 2;4:16. doi: 10.1186/s40795-018-0223-1. eCollection 2018. PMID 32153880
- [Derived] Mailey EL, Rosenkranz SK, Ablah E, Swank A, Casey K. Effects of an Intervention to Reduce Sitting at Work on Arousal, Fatigue, and Mood Among Sedentary Female Employees: A Parallel-Group Randomized Trial. J Occup Environ Med. 2017 Dec;59(12):1166-1171. doi: 10.1097/JOM.0000000000001131. PMID 28816735
- [Derived] Mailey EL, Rosenkranz SK, Casey K, Swank A. Comparing the effects of two different break strategies on occupational sedentary behavior in a real world setting: A randomized trial. Prev Med Rep. 2016 Aug 9;4:423-8. doi: 10.1016/j.pmedr.2016.08.010. eCollection 2016 Dec. PMID 27583200